CLINICAL TRIAL: NCT02681861
Title: A Phase 1 Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP6294 Administered Intravenously or Subcutaneously in Healthy Young Male and Female Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP6294 Administered Intravenously or Subcutaneously in Healthy Young Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 6294-CL-0001; 2014-003451-59 (EudraCT Number)
Record Dates: First submitted 2016-01-21; First posted 2016-02-15 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP6294
Keywords: Pharmacodynamics; Pharmacokinetics; ASP6294; Maximum tolerated dose; Healthy subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1: ASP6294 Single Ascending Intravenous Doses (Experimental): A dose escalation design will be implemented. Successive cohorts of patients (8 participants/cohort) will each be started on a fixed dose of ASP6294 or Placebo intravenously. If no dose limiting toxicities are observed escalation to the next higher dose is planned approximately every 3 weeks. Within the planned dose range, a dose lower than the next planned dose may be tested, or a dose level may be repeated, depending on emerging safety, tolerability and/or other relevant data, such as available pharmacokinetic and pharmacodynamic data of previous dose levels.
  Interventions: Drug: ASP6294 Intravenous; Drug: Placebo Intravenous
- Part 2: ASP6294 Single Ascending Subcutaneous Doses (Experimental): A dose escalation design will be implemented. Successive cohorts of patients (8 participants/cohort) will each be started on a fixed dose of ASP6294 or Placebo subcutaneously. The subcutaneous cohorts may be done in parallel with part 1, using doses which have been proven to be safe and tolerable. Within the planned dose range, a dose lower than the next planned dose may be tested, or a dose level may be repeated, depending on emerging safety, tolerability and/or other relevant data, such as available pharmacokinetic and pharmacodynamic data of previous dose levels.
  Interventions: Drug: ASP6294 Subcutaneous; Drug: Placebo Subcutaneous

INTERVENTIONS:
Drug: ASP6294 Intravenous — Intravenous (IV)
  Arms: Part 1: ASP6294 Single Ascending Intravenous Doses
Drug: ASP6294 Subcutaneous — Subcutaneous (SC)
  Arms: Part 2: ASP6294 Single Ascending Subcutaneous Doses
Drug: Placebo Intravenous — Intravenous (IV)
  Arms: Part 1: ASP6294 Single Ascending Intravenous Doses
Drug: Placebo Subcutaneous — Subcutaneous (SC)
  Arms: Part 2: ASP6294 Single Ascending Subcutaneous Doses

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single ascending intravenous doses and single subcutaneous (sc) doses of ASP6294 in healthy young male and female subjects.

This study will also evaluate the pharmacokinetics (pk) of single ascending intravenous doses and single ascending sc doses of ASP6294; determine the effect of ASP6294 administered intravenously and sc on the serum levels of circulating total Nerve Growth Factor (NGF); explore a potential gender difference in safety, tolerability and pk of single intravenous dose and single sc doses administrations of ASP6294 as well as determine the maximum tolerated dose (MTD) of single intravenous doses and single sc doses of ASP6294.

Part 2 will also evaluate the relative bioavailability of ASP6294 when administered sc.

DETAILED DESCRIPTION:
The study consists of two parts: Part 1 (ascending intravenous dose) and Part 2 (ascending subcutaneous dose). Subjects will participate in either Part 1 or Part 2. Subjects in Part 1 and Part 2 will have a residential period of 6 days followed by outpatient visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index range of 18.5 - 30.0 kg/m2, inclusive, and the subject weighs at least 50 kg (at screening).
* Female subject must either:

  * Be of non-childbearing potential: Post-menopausal (defined as at least 1 year without any menses) prior to screening, or Documented surgically sterile
  * Or, if of childbearing potential: Agree not to try to become pregnant during the study and for 120 days after final study drug administration; Must have a negative pregnancy test at screening and day -1; And, if heterosexually active, agree to consistently use 2 forms of birth control starting at screening and throughout the clinical study period and for 120 days after final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the clinical study period, and for 120 days after final study drug administration.
* Female subject must not donate ova starting at screening and throughout the clinical study period, and for 120 days after final study drug administration.
* Male subject and their female spouse/partner who are of childbearing potential must be using a highly effective form of birth control† in combination with a barrier method starting at screening and throughout the clinical study period and for 120 days after final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the clinical study period and for 120 days after final study drug administration.
* Subject agrees not to participate in another interventional study during participation in the present study, defined as signing the informed consent form until completion of the last study visit.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months prior to screening assessment or breast feeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP6294 or any components of the formulation used.
* Subject has been exposed to a biological drug within the last 6 months prior to screening.
* Subject has a history of allergic or anaphylactic reaction to a biological drug.
* Subject has been diagnosed with osteoarthritis (OA) or has a history of rapidly progressive OA.
* Subject has any of the liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, gamma glutamyl transferase, total bilirubin [TBL]) above the upper limit of normal (ULN) at day-1. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic (including orthostatic hypotension and autonomic neuropathy), dermatologic, psychiatric, renal and/or other major disease or malignancy, as judged by the investigator.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to day -1 (admission day).
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, ECG and protocol-defined clinical laboratory tests at screening or day -1.
* Subject has a mean pulse < 40 or > 90 beats per minute; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (vital sign measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) at screening and day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate measurement can be taken.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) of > 430 ms for males and > 450 ms for females at screening and day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken (admission day).
* Subject uses any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g. St. John's Wort) in the 2 weeks prior to study drug administration, except for occasional use of paracetamol (up to 2 g/day) or the use of contraceptives or hormone replacement therapy.
* Subject has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the clinical unit.
* Subject has a history of drinking more than 21 units (male subjects) or 14 units (female subjects) of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the clinical unit or the subject tests positive for alcohol or drugs of abuse at screening or day-1 (amphetamines, barbiturates, benzodiazepines, tetrahydrocannabinoids, cocaine, and opiates).
* Subject uses any drugs of abuse within 3 months prior to admission to the clinical unit.
* Subject uses any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to admission to the clinical unit regularly.
* Subject has experienced significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission to the clinical unit.
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies, hepatitis B core antibodies, or antibodies to human immunodeficiency virus types 1 and 2.
* Subject participated in any clinical study or has been treated with any investigational drugs within 3 months prior to screening.
* Subject has any condition which, in the investigator's opinion, makes the subject unsuitable for study participation, such as phobias for intravenous or subcutaneous needles/injections.
* Subject is an employee of the Astellas Group or a contract research organization.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety of ASP6294 as assessed by Nature, frequency and severity of Adverse Events (AEs) | Up to 120 Days
Safety of ASP6294 as assessed by Vital signs | Up to 120 Days
  Vital signs include blood pressure, pulse and oral body temperature
Safety of ASP6294 as assessed by Neurological examination | Up to 120 Days
  Neurological Assessment will be measured on a scale for the following Neurological examinations: Gait; Coordination; Speech; Cranial Nerves; Sensations; Muscle Strength; Muscle Tone; Muscle Movement and Reflexes and will be rated as "Normal" or "Abnormal".
Safety of ASP6294 as assessed by laboratory tests | Up to 120 Days
  Laboratory tests include hematology, biochemistry and urinalysis
Safety of ASP6294 as assessed by routine 12-lead Electrocardiogram (ECG) | Up to 120 Days
Safety of ASP6294 as assessed by continuous cardiac monitoring (Holter ECG) (part 1 only) | Days 1 and 2
  ECGs are to be collected using a 12-lead ECG continuous monitoring and recording system.
Safety of ASP6294 as assessed by Sensory assessments | Up to 120 Days
  Sensory Assessment will be measured on a scale for Lower Limbs and Hands. The following categories: Touch Pressure; Pinprick; Vibration and Joint Position will be rated as Normal (=0 points), Decreased (= 1 point) or Absent (=2 points). A total score for the left and right side of lower limbs and hands will be calculated.

SECONDARY OUTCOMES:
Pharmacokinetics of ASP6294: AUClast | Up to 120 Days
  Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast)
Pharmacokinetics of ASP6294: AUC168h | Up to 120 Days
  Area under the concentration-time curve from the time of dosing to 168 hours postdose (AUC168h)
Pharmacokinetics of ASP6294: AUCinf | Up to 120 Days
  Area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf)
Pharmacokinetics of ASP6294: Cmax | Up to 120 Days
  Maximum concentration (Cmax)
Pharmacokinetics of ASP6294: CL (part 1 only) | Up to 120 Days
  Total systemic clearance after intravenous dosing (CL)
Pharmacokinetics of ASP6294: CL/F (part 2 only) | Up to 120 Days
  Apparent total systemic clearance after extravascular dosing (CL/F)
Pharmacokinetics of ASP6294: λz | Up to 120 Days
  Terminal elimination rate constant (λz)
Pharmacokinetics of ASP6294: MRT | Up to 120 Days
  Mean residence time (MRT)
Pharmacokinetics of ASP6294: tmax | Up to 120 Days
  Time of maximum concentration (tmax)
Pharmacokinetics of ASP6294: t1/2 | Up to 120 Days
  Terminal elimination half-life (t1/2)
Pharmacokinetics of ASP6294: Vss (part 1 only) | Up to 120 Days
  Volume of distribution at steady state determined after intravenous dosing (Vss)
Pharmacokinetics of ASP6294: Vz (part 1 only) | Up to 120 Days
  Volume of distribution during terminal elimination phase after intravenous dosing (Vz)
Pharmacokinetics of ASP6294: Vz/F (part 2 only) | Up to 120 Days
  Apparent volume of distribution during the terminal elimination phase after extravascular dosing (Vz/F)
Pharmacodynamics of ASP6294 Nerve growth factor (NGF) total serum concentration: Cmax | Up to 120 Days
Pharmacodynamics of ASP6294 NGF total serum concentration: tmax | Up to 120 Days

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Site GB44001, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided